CLINICAL TRIAL: NCT06779695
Title: Prediction of Systemic Thromboembolism and Bleeding in Atrial Fibrillation Patients With Factor Xa Inhibitor (Apixaban, Rivaroxaban) by Echocardiographic Parameters: Prospective Observational Study (AF-ECHO Study)
Status: Active, not recruiting | Type: Observational
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Korea University Ansan Hospital (Other); Mediplex Sejong Hospital (Unknown); Chungnam National University Hospital (Other); Chonnam National University Hospital (Other); Kyung Hee University Hospital at Gangdong (Other); Kyungpook National University Hospital (Other); Korea University Guro Hospital (Other); InjeUniversityIlsanPaikHospital (Unknown); Wonkwang University Hospital (Other); Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Mi Park, M.D. Ph.D., Professor, Korea University Anam Hospital
Other Study IDs: 2024AN0119
Record Dates: First submitted 2025-01-13; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Apixaban,; Rivaroxaban
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic AF who have started taking Factor Xa inhibitors.: Patients aged 19 and over with chronic atrial fibrillation who have started taking Factor Xa inhibitors (Apixaban, Rivaroxaban), within the last 12 months and have obtained an echocardiography image that can be analyzed within 3 months.

SUMMARY:
Patients taking Factor Xa inhibitors (Apixaban, Rivaroxaban) in atrial fibrillation will be conducted a follow-up investigation on systemic embolism and bleeding events.

DETAILED DESCRIPTION:
This study aims to evaluate 1) the efficacy and safety of Factor Xa inhibitors (Apixaban, Rivaroxaban) in atrial fibrillation patients who meet the inclusion criteria, and 2) the relationship between systemic embolism and bleeding by tracking and analyzing echocardiographic data, with the goal of developing an AF-ECHO NOAC Score to predict these events. Additionally, we aim to create a predictive model for thromboembolic and bleeding events by observing the occurrence and progression of mitral and tricuspid regurgitation due to atrial remodeling and annular dilation in atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria

1. Male and female patients aged 19 years or older with chronic atrial fibrillation, accompanied by at least one of the following conditions:

   ① Heart failure

   ② 2. Myocardial infarction (more than 3 months post-event)

   ③ 3. Angina (if PCI was performed, more than 3 months post-procedure)

   ④ 4. Hypertension

   ⑤ 5. Diabetes mellitus
2. Patients who started taking Factor Xa inhibitors (Apixaban, Rivaroxaban) within the last 12 months and have echocardiographic images taken within 3 months of that time, which are available for analysis.
3. Patients who are starting treatment with Factor Xa inhibitors. (Apixaban, Rivaroxaban)
4. Individuals who have voluntarily provided written consent to participate in this clinical trial.

Exclusion Criteria

1. Patients with creatinine clearance (CCr) less than 15 ml/min.
2. Patients with moderate to severe mitral stenosis.
3. Patients who have undergone mechanical valve replacement
4. Patients with a history of clinically significant alcohol or drug abuse.
5. Patients whom the investigator deems legally or mentally unsuitable for participation in the clinical trial, or those who do not consent to participate in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atrial fibrillation patients from 11 institutions who are taking or starting Factor Xa inhibitors (Apixaban, Rivaroxaban)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-04-21 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome MeasureIdentification of risk factors for systemic embolism and bleeding through echocardiography in atrial fibrillation patients taking Factor Xa inhibitors (Apixaban, Rivaroxaban) | From enrollment to the end of treatment at 60 months.
  We aim to retrospectively and prospectively assess the risk of systemic embolism and bleeding in Korean patients with atrial fibrillation who are taking oral anticoagulants, specifically Factor Xa inhibitors (Apixaban, Rivaroxaban). Additionally, we will evaluate echocardiographic parameters such as ventricular and atrial function, as well as valvular regurgitation, which are expected to influence the occurrence of embolism and bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Na Kim, M.D., Ph.D., Study Chair — Korea University Anam Hospital; Dong-Hyuk Cho, PhD, Study Chair — Korea University Anam Hospital; So Ree Kim, PhD, Study Chair — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yao Y, Zhang Z, Xue J, Chen Z, Zhou Y, Luo W, Ye F, Wang J, Long D. Echocardiographic Mitral Annular Calcification is Associated With Atrial Fibrillation Recurrence After Catheter Ablation. Am J Cardiol. 2023 Apr 15;193:55-60. doi: 10.1016/j.amjcard.2023.01.054. Epub 2023 Mar 3. PMID 36871530
- [Result] Lu ML, Gupta S, Romero-Corral A, Matejkova M, De Venecia T, Obasare E, Bhalla V, Pressman GS. Cardiac Calcifications on Echocardiography Are Associated with Mortality and Stroke. J Am Soc Echocardiogr. 2016 Dec;29(12):1171-1178. doi: 10.1016/j.echo.2016.08.020. Epub 2016 Oct 11. PMID 27742243
- [Result] Liao JN, Chao TF, Kuo JY, Sung KT, Tsai JP, Lo CI, Lai YH, Su CH, Hung CL, Yeh HI. Global Left Atrial Longitudinal Strain Using 3-Beat Method Improves Risk Prediction of Stroke Over Conventional Echocardiography in Atrial Fibrillation. Circ Cardiovasc Imaging. 2020 Aug;13(8):e010287. doi: 10.1161/CIRCIMAGING.119.010287. Epub 2020 Aug 13. PMID 32787500
- [Result] Thomas KL, Jackson LR 2nd, Shrader P, Ansell J, Fonarow GC, Gersh B, Kowey PR, Mahaffey KW, Singer DE, Thomas L, Piccini JP, Peterson ED. Prevalence, Characteristics, and Outcomes of Valvular Heart Disease in Patients With Atrial Fibrillation: Insights From the ORBIT-AF (Outcomes Registry for Better Informed Treatment for Atrial Fibrillation). J Am Heart Assoc. 2017 Dec 22;6(12):e006475. doi: 10.1161/JAHA.117.006475. PMID 29273635
- [Result] Qamar A, Vaduganathan M, Greenberger NJ, Giugliano RP. Oral Anticoagulation in Patients With Liver Disease. J Am Coll Cardiol. 2018 May 15;71(19):2162-2175. doi: 10.1016/j.jacc.2018.03.023. PMID 29747837
- [Result] Lee HF, Chan YH, Chang SH, Tu HT, Chen SW, Yeh YH, Wu LS, Kuo CF, Kuo CT, See LC. Effectiveness and Safety of Non-Vitamin K Antagonist Oral Anticoagulant and Warfarin in Cirrhotic Patients With Nonvalvular Atrial Fibrillation. J Am Heart Assoc. 2019 Mar 5;8(5):e011112. doi: 10.1161/JAHA.118.011112. PMID 30834802
- [Result] Chatterjee NA, Shah RV, Murthy VL, Praestgaard A, Shah SJ, Ventetuolo CE, Barr RG, Kronmal R, Lima JA, Bluemke DA, Jerosch-Herold M, Alonso A, Kawut SM. Right Ventricular Structure and Function Are Associated With Incident Atrial Fibrillation: MESA-RV Study (Multi-Ethnic Study of Atherosclerosis-Right Ventricle). Circ Arrhythm Electrophysiol. 2017 Jan;10(1):e004738. doi: 10.1161/CIRCEP.116.004738. PMID 28082528
- [Result] Rutherford OW, Jonasson C, Ghanima W, Holst R, Halvorsen S. New score for assessing bleeding risk in patients with atrial fibrillation treated with NOACs. Open Heart. 2018 Dec 9;5(2):e000931. doi: 10.1136/openhrt-2018-000931. eCollection 2018. PMID 30613418